CLINICAL TRIAL: NCT00000703
Title: Chemotherapy and Azidothymidine, With or Without Radiotherapy, for High Grade Lymphoma in AIDS-Risk Group Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 008; 10984 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: Vincristine; Lymphoma; Methotrexate; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Drug Therapy, Combination; Combined Modality Therapy; Acquired Immunodeficiency Syndrome; Antineoplastic Agents, Combined; Zidovudine; Bleomycin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Lymphoma; Acquired Immunodeficiency Syndrome | interventions — Bleomycin; Vincristine; Doxorubicin; Cyclophosphamide; Allopurinol; Methotrexate; Cytarabine; Leucovorin; Zidovudine; Dexamethasone

INTERVENTIONS:
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Cyclophosphamide
Drug: Allopurinol
Drug: Methotrexate
Drug: Cytarabine
Drug: Leucovorin calcium
Drug: Zidovudine
Drug: Dexamethasone

SUMMARY:
To determine the safety and effectiveness of a combination chemotherapy-radiation-zidovudine (AZT) treatment for patients with peripheral lymphoma.

Other chemotherapies have been tried in patients with AIDS related lymphomas, but the results have not been satisfactory. This study will show whether the combination of chemotherapy, radiation, and AZT is more effective and less toxic than previously used treatments.

DETAILED DESCRIPTION:
Other chemotherapies have been tried in patients with AIDS related lymphomas, but the results have not been satisfactory. This study will show whether the combination of chemotherapy, radiation, and AZT is more effective and less toxic than previously used treatments.

All patients will receive combination chemotherapy and AZT. The combination chemotherapy will be repeated every 3 to 4 weeks for a maximum total of 6 cycles. Each cycle will consist of doxorubicin, bleomycin, cyclophosphamide, and vincristine on day 1, dexamethasone on days 1-5, and methotrexate on day 15. Patients with meningeal or bone marrow disease will receive radiation and intrathecal cytarabine (ARA-C) while those without will receive ARA-C without radiation. Patients with documented lymphomas in the central nervous system at initial workup will start radiation as soon as possible and intrathecal ARA-C (t.i.w. until cerebrospinal fluid is clear then every month for 1 year); patients with normal lumbar puncture, brain scan, and bone marrow at first diagnosis will begin radiation on day 1 of cycle 3 of chemotherapy. Lumbar punctures for evaluation will be done four times during the first cycle, on days 1, 8, 21, and 28. AZT will be administered every 4 hours, 7 days a week, beginning at the completion of combined chemotherapy, once the patient has achieved a complete remission of the lymphoma, and continuing for 1 year.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Ibuprofen.
* Standard antiemetic agents.
* Ganciclovir therapy for sight- or life-threatening Cytomegalovirus infection.
* Zidovudine and methotrexate may be resumed during ganciclovir maintenance phase.

Exclusion Criteria

Co-existing Condition:

The following patients will be excluded from the study:

* Patients with recurrent infection that may interfere with the planned protocol.
* Patients with a second active tumor other than nonmelanomatous skin cancer or Kaposi's sarcoma.
* Patients with stage IE primary central nervous system lymphoma.

Concurrent Medication:

Excluded:

* Corticosteroids.
* Aspirin.
* Acetaminophen.
* Nonsteroidal anti-inflammatory drugs, except ibuprofen.
* Chemotherapy for infection associated with neutropenia.
* Zidovudine (AZT) for infection associated with neutropenia.
* Investigational therapies, except ganciclovir therapy for sight- or life-threatening cytomegalovirus infection.
* AZT and methotrexate will be suspended during induction therapy with ganciclovir.

The following patients will be excluded from the study:

* Patients with recurrent infection that may interfere with the planned protocol.
* Patients with a second active tumor other than nonmelanomatous skin cancer or Kaposi's sarcoma.
* Patients with stage IE primary central nervous system lymphoma.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Excluded within 2 weeks of study entry:
* Immunomodulating agents.
* Antiretroviral therapy prior to diagnosis of lymphoma.

Patients must demonstrate the following clinical and laboratory findings:

* Any stage of the disease, including stage I.
* Newly diagnosed, previously untreated high-grade lymphoma.
* Presence of measurable tumor parameter(s).
* Adequate hepatic, renal, and bone marrow function.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Study Completion 1990-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levine A, Study Chair
Locations (14):
- United States (14):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Saag MS, Emini EA, Laskin OL, Douglas J, Lapidus WI, Schleif WA, Whitley RJ, Hildebrand C, Byrnes VW, Kappes JC, et al. A short-term clinical evaluation of L-697,661, a non-nucleoside inhibitor of HIV-1 reverse transcriptase. L-697,661 Working Group. N Engl J Med. 1993 Oct 7;329(15):1065-72. doi: 10.1056/NEJM199310073291502. PMID 7690462
- [Background] Levine AM, Wernz JC, Kaplan L, Rodman N, Cohen P, Metroka C, Bennett JM, Rarick MU, Walsh C, Kahn J, et al. Low-dose chemotherapy with central nervous system prophylaxis and zidovudine maintenance in AIDS-related lymphoma. A prospective multi-institutional trial. JAMA. 1991 Jul 3;266(1):84-8. PMID 1710673
- [Background] ICDB/89653727. Levine AM, et al. Low dose chemotherapy with CNS prophylaxis and zidovudine (AZT) maintenance for aids-related lymphoma: preliminary results of a multi-institutional study. Proc Annu Meet Am Soc Clin Oncol. 1989 8:A18